CLINICAL TRIAL: NCT00875394
Title: A Multicenter, Randomized, Open-label Study to Assess the Efficacy and Safety of Sitagliptin Added to the Regimen of Patients With T2 DM With Inadequate Glycemic Control on Metformin
Brief Title: Study to Assess the Efficacy and Safety of Sitagliptin Added to the Regimen of Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin (0431-189)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-189; 2009_571
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): sitagliptin + metformin
  Interventions: Drug: sitagliptin phosphate; Drug: Comparator: metformin
- 2 (Active Comparator): metformin + any other oral antidiabetic drug
  Interventions: Drug: Comparator: metformin; Drug: Comparator: Antidiabetic Standard of Care
- 3 (Active Comparator): metformin
  Interventions: Drug: Comparator: metformin

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin 100 mg Once a day (QD) for 24 weeks
  Other Names: sitagliptin
  Arms: 1
Drug: Comparator: metformin — metformin 850 mg Twice a day (BID) for 24 weeks
  Other Names: metformin
  Arms: 1; 2
Drug: Comparator: metformin — metformin 500 mg Three times a day (TID) to 850 mg Twice a day (BID), for 24 weeks
  Other Names: metformin
  Arms: 3
Drug: Comparator: Antidiabetic Standard of Care — Patient can take any oral antidiabetic drug (other than metformin)
  Arms: 2

SUMMARY:
After 24 weeks of treatment, to assess the A1C-lowering efficacy of sitagliptin 100 mg once daily added to the regimen of patients with inadequate glycemic control on metformin monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patient Has Type 2 Diabetes Mellitus
* Patient Is 30-78 Years Of Age On The Day Of Signing Informed Consent
* Patient Is Currently On Metformin Therapy (1500 Mg/Day)
* Patient Is A Male Or A Female Who Is Unlikely To Conceive, As Indicated By At Least One Yes Answer To The Following Questions: A) Patient Is A Male. B) Patient Is A Surgically Sterilized Female. C) Patient Is A Postmenopausal Female 45 Years Of Age With >2 Years Since Last Menses. D) Patient Is A Non-Sterilized Premenopausal Female And Agrees To Use An Adequate Method Of Contraception To Prevent Pregnancy Throughout The Study Starting With Visit 1 And For 14 Days After The Last Dose Of Study Medication
* Patient Understands The Study Procedures, The Alternative Treatments Available, The Risks Involved In The Study And Voluntarily Agrees To Participate By Giving Written Informed Consent
* Patient Has An A1c of 6.5 % - 11.0%

Exclusion Criteria:

* Patient Has A History Of Type 1 Diabetes Mellitus Or History Of Ketoacidosis

Ages: 30 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2008-06-27 (Actual); Study Completion 2008-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in Principal Investigator's private practice, in Mexico City.
  First Patient Entered: 15 Feb 2007. Last Patient's Last Visit: 27 Jun 2008
Pre-assignment Details: Patients 30 to 78 years of age with inadequate glycemic control (Glycosylated hemoglobin A1C (A1C) 6.5 to 11%) on diet/exercise and metformin dosed at ≥1500 mg per day patients were to receive either sitagliptin added to ongoing metformin or "standard care" added to ongoing metformin.
Groups:
- Sitagliptin + Metformin: Patients administered sitagliptin and metformin
- Metformin + Any Non-DPP-4i Oral Antidiabetic Drug; Metformin Alone: Patients in the 'standard care' group were to receive continued treatment with metformin and usual care per practice but not to be treated with sitagliptin or another Dipeptidyl peptidase 4 inhibitor (DPP-4i). As prespecified in the protocol, no efficacy was to be assessed for patients receiving "standard care".
Period: Overall Study
Arm/Group | Sitagliptin + Metformin | Metformin + Any Non-DPP-4i Oral Antidiabetic Drug | Metformin Alone
Started | 36 | 23 | 9
Completed | 36 | 23 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin + Metformin | Metformin + Any Non-DPP-4i Oral Antidiabetic Drug | Metformin Alone | Total
Number analyzed (Participants) | 36 | 23 | 9 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (9.8) | 56.0 (8.5) | 53.3 (11.7) | 54.69 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 6 | 50
  Male | 11 | 4 | 3 | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 29.0 (4.5) | 28.8 (5.1) | 28.3 (5.2) | 28.84 (4.74)
Glycosylated Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 8.8 (1.5) | 8.0 (1.8) | 8.2 (1.1) | 8.47 (1.61)
Time since diagnosis of diabetes [Mean (Standard Deviation); unit: Years] | 8.9 (7.1) | 6.8 (8.5) | 10.9 (7.7) | 8.43 (7.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1C (A1C) at Week 24
Description: Week 24 A1C minus baseline (Week 0) A1C. The unit for A1C is "percent". Thus, this measure represents a difference of percent values.
Time Frame: Baseline and 24 weeks
Population: Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.
Arm/Group | Sitagliptin + Metformin | Metformin + Any Non-DPP-4i Oral Antidiabetic Drug | Metformin Alone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sitagliptin + Metformin | Metformin + Any Non-DPP-4i Oral Antidiabetic Drug | Metformin Alone
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/23 | 0/9
Other Adverse Events (participants affected / at risk) | 0/36 | 1/23 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin + Metformin (N=36) | Metformin + Any Non-DPP-4i Oral Antidiabetic Drug (N=23) | Metformin Alone (N=9)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
A limited number of participants were recruited into this open-label study. This study was conducted at a single site.

Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.